CLINICAL TRIAL: NCT06618963
Title: Effect of Omalizumab in the Skin of Food Allergy Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RO-IIS-1660
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-09

CONDITIONS: Food Allergy; Food Allergy in Children
Keywords: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: 30 subjects with food allergy 10 subjects without food allergy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Food Allergy (Active Comparator): This group will receive 4 months of Omalizumab treatment, and undergo regular skin barrier assessments.
  Interventions: Drug: Omalizumab Injection
- Participants without Food Allergy (No Intervention): This group will undergo skin barrier assessment.

INTERVENTIONS:
Drug: Omalizumab Injection — Omalizumab is a monoclonal antibody FDA-approved for treatment of food allergy.
  Other Names: Xolair
  Arms: Participants with Food Allergy

SUMMARY:
The goal of this interventional study is to evaluate whether skin barrier abnormalities occur in subjects with a food allergy, as determined by positive oral food challenge (OFC). The main question it aims to answer is whether these skin barrier abnormalities can be reversed by omalizumab.

If there is a comparison group: Researchers will compare non-food allergic participants (who do not receive omalizumab) to see if they experience skin barrier abnormalities.

All food allergic participants will receive 4 months of Omalizumab treatment as well as two Oral Food Challenges. Participants will all undergo skin barrier assessments.

DETAILED DESCRIPTION:
This is a phase IV open-label interventional pilot study of 30 patients enrolled at National Jewish Health to examine skin barrier function and response to OFC in patients with FA before and after 4 months of treatment with omalizumab. If enrollment is insufficient at National Jewish, Children's Hospital Colorado or another similarly qualified site will be used as a back-up site. Efficacy assessment will be assessed by the ability of Omalizumab to reduce clinical response to OFC. The safety of omalizumab will be concomitantly recorded. Specifically, we will:

1. Examine TEWL, STS lipidomics, metabolomics, cytokines, and proteomics in 30 patients with a history of IgE-mediated reaction to 1 or more foods assessed by sensitization food extracts using skin prick tests, serum IgE to specific foods and/or relevant component proteins, and an IgE-mediated clinical reaction to a food on OFC.
2. Confirm the diagnosis of IgE-mediated FA in all patients with a positive OFC.
3. Treat all 30 patients with omalizumab for 4 months
4. Repeat OFC after 4 months of omalizumab therapy.
5. To analyze TEWL, STS Lipidomics, metabolomics, proteomics, and cytokines in all 30 patients who were treated with omalizumab and completed the end of study OFC.

Sample size will be 30 completed subjects. Enrollment will occur over the course of 16 months, with 2-4 participants enrolling each month. Up to ten healthy control subjects will also be enrolled for skin tape strip analysis and TEWL as a comparator group to the FA group.

All participants will have an initial screening visit where their clinical history of having an IgE-mediated reaction to specified food(s) will be elucidated, along with review of relevant skin prick test (SPT), food-specific IgE values, and Total IgE. If these values were not obtained within the last 12 months, SPT, sIgE, and/or Total IgE will be performed at screening. All food-allergic participants will undergo an open Screening OFC to one of their food allergens. For continuation in the study, the participant must experience dose-limiting symptoms consistent with an IgE-mediated reaction, at or before 444mg of food protein cumulatively. If they have a negative OFC, additional screening OFCs may be performed to any eligible food. STS and TEWL measurements will be performed prior to the first dose, as well as before the second and third doses. If/when the participant has dose-limiting symptoms, STS and TEWL will be stopped immediately.

All food-allergic participants will receive omalizumab for 4 months. All injections will be administered by a research nurse on the clinical research unit. At the midway point of the study (2 months after the first omalizumab injection), the participant will have STS and TEWL measurements performed.

After 4 months of omalizumab administration, an end of study OFC will be performed to the same food that was positive at the screening OFC to assess treatment effect, along with analysis of the STS and TEWL.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or parent/legal guardian must be able to understand and provide informed consent and/or assent, as applicable.
* Male or female, 1-55 years old at screening.
* Total IgE level within 1 year of screening and weight at screening visit that together result in an eligible omalizumab dose according to the dosing table for FA (Appendix 8).
* Participant must meet the following clinical FA criteria: Food sensitization to peanut, hen's egg, a tree nut, sesame seed, cow's milk, wheat, or soy, within 1 year of screening AND experience dose-limiting, IgE mediated symptoms at or before 444mg of food protein cumulatively during screening OFC to peanut, hen's egg, a tree nut, sesame seed, cow's milk, wheat, or soy.
* If female of child-bearing potential, must have a negative urine or serum pregnancy test. If participating as a healthy control, self-report of pregnancy status is acceptable.
* For women of child-bearing potential, must agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods (barrier methods or oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy) during the treatment period and for 60 days after the last dose of study drug.
* Be willing to be trained on the proper use of an epinephrine autoinjector and be willing to always have epinephrine autoinjector immediately available for the duration of the study.

Exclusion Criteria:

* Inability or unwillingness of a participant and/or parent/legal guardian to give written informed consent and/or assent or comply with the study protocol.
* Clinically significant laboratory abnormalities at Screening.
* Sensitivity or suspected/known allergy to any ingredients (including excipients) of the active OFC material (other than the study food), or drugs related to omalizumab (e.g., monoclonal antibodies, polyclonal gamma globulin).
* Poorly controlled AD at Screening, per the PI's discretion.
* Poorly controlled or severe asthma/wheezing at Screening
* History of severe anaphylaxis (defined as neurological compromise or requiring intubation) to a study food that is to be used for qualifying OFC in this study.
* Treatment with oral, intramuscular (IM), or intravenous (IV) steroids of more than two days for an indication other than asthma/wheezing within 30 days of Screening.
* Currently receiving oral, IM, or IV corticosteroids, tricyclic antidepressants, or β-blockers (oral or topical).
* Past or current history of cancer, or currently being investigated for possible cancer.
* Previous adverse reaction to omalizumab.
* Past or current history of any immunotherapy to the OFC food (e.g., oral immunotherapy [OIT], sublingual immunotherapy [SLIT], or patch/epicutaneous immunotherapy [EPIT)] within 4 months of Screening.
* Treatment with monoclonal antibody therapy, such as omalizumab (Xolair®), dupilumab (Dupixent®), benralizumab (Fasenra™), mepolizumab (Nucala®), reslizumab (Cinqair®), or other immunomodulatory therapy within four months of Screening.
* Currently on "build-up phase" of inhalant allergen immunotherapy (i.e., has not reached maintenance dosing). Individuals tolerating maintenance allergen immunotherapy can be enrolled.
* Inability to discontinue antihistamines for the minimum wash-out periods required for SPTs or OFCs
* Current participation in another therapeutic or interventional clinical trial or participation within 90 days of Screening.
* Use of investigational drugs within 24 weeks of Screening.
* Pregnant or breastfeeding or intending to become pregnant during the study or within 60 days after the last dose of omalizumab.
* Have any skin disease other than AD that might compromise the stratum corneum barrier.
* History of serious life-threatening reaction to tape or adhesives.
* Healthy Control Participants (non-Food Allergy participants) may not have atopic dermatitis, autoimmune, or other conditions which, in the opinion of the PI, could confound the results of the study assessments or samples.

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lipidomic analysis | 5 months
  Lipid measurements from Skin Tape Strips (STS), as detected at respective m/z from mass spectrometry
Metabolomic analysis | 5 months
  Metabolomics from STS, evaluated as a relative signal proportion of metabolites against the sum of all signals in the samples
Proteomic analysis | 5 months
  Proteomics from STS, comparison of global protein expression before vs after omalizumab treatment
Cytokine analysis | 5 months
  Cytokine levels from STS measured using preconfigured multiplex assays normalized to the total protein in each sample. Cytokines that will be measured: IL-1a, IL-1b, IL-18, IL-6, IL-8, TARC, MDC, TSLP, IL-33, IL-4, IL-13, IL-22, IL-31, eotaxins, IL-10, IL-17A/F, IL-17C, IL-12p70, IL-23, IP-10
Measurement of Transepidermal Water Loss | 5 months
  Transepidermal Water Loss (TEWL) is measured by the loss through the skin of grams of water per square meter per hour (g/m^2/h).

SECONDARY OUTCOMES:
Measurement of Transepidermal Water Loss in non Food-Allergic Subjects | 5 months
  Transepidermal Water Loss (TEWL), grams water per square meter per hour (g/m^2/h)
Lipidomic analysis in non Food-Allergic participants | 5 months
  Lipid measurements from Skin Tape Strips (STS), as detected at respective m/z from mass spectrometry
Metabolomic analysis in non Food-Allergic Participants | 5 months
  Metabolomics from STS, evaluated as a relative signal proportion of metabolites against the sum of all signals in the samples
Proteomic analysis in non Food-Allergic Participants | 5 months
  Proteomics from STS, baseline expression levels of proteins found in non-allergic skin tapes.
Cytokine analysis | 5 months
  Cytokine levels from STS from non-Food Allergic participants, measured using preconfigured multiplex assays normalized to the total protein in each sample. Cytokines that will be measured: IL-1a, IL-1b, IL-18, IL-6, IL-8, TARC, MDC, TSLP, IL-33, IL-4, IL-13, IL-22, IL-31, eotaxins, IL-10, IL-17A/F, IL-17C, IL-12p70, IL-23, IP-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No